CLINICAL TRIAL: NCT00890032
Title: Recurrent GBM Stem Cell Tumor Amplified RNA Immunotherapy Trial
Brief Title: Vaccine Therapy in Treating Patients Undergoing Surgery for Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Sampson (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Sampson, Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006677; R01CA135272 (NIH); P30CA014236 (NIH); CDR0000630701 (Other: NCI)
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Central Nervous System Neoplasm
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult astrocytoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BTSC mRNA-loaded DCs (Experimental): BTSC mRNA-loaded DCs administered intradermally weekly for first 3 vaccines, then monthly until progression or withdrawal.
  Interventions: Biological: BTSC mRNA-loaded DCs

INTERVENTIONS:
Biological: BTSC mRNA-loaded DCs — An escalating total dose of BTSC mRNA-loaded DCs (2x10^6, 5x10^6, and 2x10^7 per vaccination) will be evaluated for purpose of establishing a maximum tolerated dose (MTD) and a dose-limiting toxicity (DLT).

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and dendritic cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy in treating patients undergoing surgery for recurrent glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility and safety of an autologous brain tumor stem cell messenger ribonucleic acid (mRNA)-loaded dendritic cell vaccine in adult patients with recurrent glioblastoma multiforme.

Secondary

* To assess humoral and cellular immune responses to vaccination.
* To compare the proportion of vaccinated patients alive at 6 months from the time of surgery for recurrent tumor with matched historical cohorts.

OUTLINE: Patients undergo surgical resection of tumor. Tumor tissue samples are collected to isolate brain tumor stem cells (BTSCs) and for extraction and amplification of BTSC-specific mRNA. Within 4 weeks after surgical resection, patients undergo leukapheresis over 4 hours to generate dendritic cells (DCs). Patients also undergo leukapheresis at 1 week after the third vaccination and then at least every 3 months as needed for generation of additional DCs.

Patients receive autologous BTSC mRNA-loaded DC vaccine intradermally once weekly for 3 weeks and then once monthly in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* First recurrence of GBM (WHO Grade IV glioma or astrocytoma) in surgically accessible areas with prior histologic diagnosis of GBM
* No known contraindications to receiving Avastin
* Karnofsky Performance Status (KPS) of > 70%
* Radiation Therapy (RT) with ≥ 45 Gy tumor dose, completed ≥ 8 weeks prior to study entry

Exclusion Criteria:

* Contrast-enhancing tumor component crossing the midline, multi-focal tumor, or tumor dissemination (subependymal or leptomeningeal)
* Clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment
* Pregnant or need to breast feed during the study period (Negative beta-human chorionic gonadotropin (HCG) test required), or unable to maintain use of contraception while on study
* Active infection requiring treatment or an unexplained febrile (> 101.5 degrees F) illness
* Known immunosuppressive disease, autoimmune disease or human immunodeficiency virus infection, Hepatitis B or Hepatitis C
* Unstable or severe intercurrent medical conditions such as severe heart (New York Association Class 3 or 4) or lung (FEV1 < 50%) disease, uncontrolled diabetes mellitus
* Prior brachytherapy, carmustine wafer therapy, radiolabeled monoclonal antibodies, or stereotactic radiosurgery
* Prior inguinal lymph node dissection

Avastin-Specific Exclusion Criteria

Subjects meeting any of the following criteria are ineligible for study entry:

* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to enrollment
* History of stroke or transient ischemic attack within 6 months prior to enrollment
* Significant vascular disease (e.g. aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) (within 6 months prior to enrollment)
* History of hemoptysis (> or = 1/2 teaspoon of bright red blood per episode) within 28 days prior to enrollment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to enrollment
* Serious, non-healing wound, active ulcer or untreated bone fracture
* Proteinuria as defined by > +1 on urinalysis dipstick
* Known hypersensitivity to any component of Avastin
* Pregnant (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety | 12 months

SECONDARY OUTCOMES:
Humoral and cellular immune responses | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Vlahovic, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States